CLINICAL TRIAL: NCT01422603
Title: A Pilot Study of Clofarabine Pre-conditioning Prior to Full or Reduced Intensity Allogeneic Transplantation in the Treatment of High Risk Acute Myeloid Leukaemia and Myelodysplasia.
Brief Title: Clofarabine Pre-conditioning With Allogeneic Transplant for Acute Myeloid Leukaemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHM CAN0638; 2008-007043-14 (EudraCT Number)
Record Dates: First submitted 2011-08-22; First posted 2011-08-24 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Acute Myeloid Leukaemia; Myelodysplasia
Keywords: High risk; AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clofarabine and Full intensity SCT (Experimental): Cohort One: Patients suitable for full intensity conditioning will receive Clofarabine pre-conditioning followed by a Cyclophosphamide and Total Body Irradiation conditioned allogeneic stem cell transplant (SCT).
  Interventions: Drug: Clofarabine
- Clofarabine and Reduced intensity SCT (Experimental): Cohort 2: Patients not suitable for a full intensity TBI-based transplant due to age or co-morbidity will receive Clofarabine pre-conditioning followed by a reduced intensity allogeneic stem cell transplant using Fludarabine, intravenous Busulphan and Campath 1H.
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Clofarabine preconditioning (40mg/m2 daily for 5 days) prior to full intensity allogeneic stem cell transplant
  Arms: Clofarabine and Full intensity SCT
Drug: Clofarabine — Clofarabine preconditioning (40mg/m2 daily for 5 days) prior to reduced intensity allogeneic stem cell transplant
  Arms: Clofarabine and Reduced intensity SCT

SUMMARY:
This study has been designed to investigate the safety and feasibility of using a chemotherapy drug, Clofarabine, to reduce the disease burden before a donor transplant, in patients with high risk Acute Myeloid Leukaemia or Myelodysplasia (MDS). In this study Clofarabine chemotherapy will be given a few days before a reduced or full intensity donor stem cell transplant and without waiting for normal blood counts to recover. It is hoped that this approach may improve the outcome for patients with high risk AML and MDS after their transplant.

DETAILED DESCRIPTION:
This is a pilot study. Twenty patients in total will be treated in two cohorts of 10 patients each.

* Cohort One: Patients suitable for full intensity conditioning will receive Clofarabine pre-conditioning followed by a Cyclophosphamide and Total Body Irradiation conditioned allogeneic stem cell transplant.
* Cohort Two: Patients not suitable for a full intensity TBI-based transplant due to age or co-morbidity will receive Clofarabine pre-conditioning followed by a reduced intensity allogeneic stem cell transplant using Fludarabine, intravenous Busulphan and Campath 1H.

The cohorts will be recruited concurrently. It is anticipated that recruitment of the 20 subjects will be achieved in 18 months to two years.

The study will be conducted at a single centre (Southampton, UK) in the first instance.

This design allows the use of a full intensity, TBI-based transplant conditioning schedule, for younger patients able to tolerate this approach but also the use of a reduced intensity transplant conditioning schedule in older or less fit patients who may still benefit from pre-conditioning with Clofarabine followed by an allogeneic stem cell transplant. This design, therefore, does not restrict potential recruitment to the study on age or performance status alone (within the limits set by ability to tolerate intensive chemotherapy and a transplant procedure).

ELIGIBILITY:
Inclusion Criteria:

* Cytologically and immunophenotypically (or immunohistochemically) confirmed diagnosis of high risk AML or MDS
* Minimum age of 18 years
* Eligible for allogeneic stem cell transplant by local institutional guidelines
* Suitable matched-related/sibling or volunteer unrelated donor available, as determined by local institutional guidelines
* Negative pregnancy test for females of child-bearing potential within 7 days prior to the start of study treatment
* If sexually active, male and female subjects must agree that they will use an effective method of birth control throughout the active study period
* Written informed consent
* Capable of and willing to comply with scheduled visits, treatment plan and required laboratory tests
* Adequate renal and hepatic function

Exclusion Criteria:

* Psychiatric, addictive or any disorder which compromises ability to give truly informed consent for participation in this study
* Previous Allogeneic Bone Marrow or Peripheral Blood Stem Cell Transplant.
* Pregnant or lactating women. All female subjects of child-bearing potential must have a negative pregnancy test within 7 days prior to the start of treatment.
* Any current active, invasive malignancy excluding AML or MDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-02; Primary Completion 2014-05 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Treatment related mortality (TRM) | day 100 and 1 year post transplant
  Treatment related mortality (TRM) measured at day 100 and 1 year post transplant and cause of mortality

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year post transplant
Event free survival (EFS) | 1 year post transplant
Efficacy of Clofarabine as a leukaemia bulk-reducing agent prior to transplant conditioning | Within 4 weeks prior to Clofarabine and 1 to 5 days following Clofarabine
  Efficacy of Clofarabine as a leukaemia bulk-reducing agent prior to transplant conditioning as determined by pre- and post-Clofarabine bone marrow biopsy examination
Time to engraftment | by day 100 post transplant
Donor/recipient chimerism | day 30, day 100 and 1 year post transplant
Immune reconstitution parameters (T, B and NK cell subsets) | day 30, day 100 and 1 year post transplant
Duration of hospital stay | The duration of hospital stay will be measured, an expected average of 7 to 8 weeks
  Duration of in patient hospital stay for Clofarabine preconditioning chemotherapy and stem cell transplant
Incidence of acute and chronic graft versus host disease | 1 year post transplant
Grade of acute and chronic graft versus host disease | 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Deborah S Richardson, MA MB BChir MD FRCP FRCPath, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Wessex Blood and Marrow Transplant Unit, Southampton University Hospitals NHS Trust, Southampton, Hampshire, United Kingdom